CLINICAL TRIAL: NCT01770925
Title: Non-invasive Ventilation as a Post Extubation Mode for RDS: a Randomized, Cotrolled Trial to Compare n-CPAP by n- Bipap and NIPPV
Brief Title: n-CPAP Versus n-BiPAP and NIPPV for Postextubation in RDS in Preterms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ali El-Farrash, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ain shams university; riham samy (Registry Identifier: rania ali)
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- n-CPAP (Active Comparator): * The n-CPAP group will receive at extubation a single level continuous positive airway pressure of 7 cm water for at least 48 hours before weaning is commenced. If the infant is stable for the preceding 48 hours defined by having fewer than three minor apneas and no increase in oxygen requirement, weaning will be permitted.
  * CPAP will be decreased from 6 cm water by 1 cm water every 24 hours if tolerated based on the above criteria. This will be done until a pressure of 4 cm water is reached.
  * If a pressure of 4 cm water is successfully tolerated for 48 hours then time off n-CPAP will be allowed. Thereafter, no fixed weaning regime based on number of hours in a day the infant will be allowed to come off CPAP will be prescribed.
  Interventions: Device: N-CPAP
- n-BiPAP (Active Comparator): * The n-BiPAP group will receive at extubation a mean airway pressure of 7 cm water (positive end expiratory pressure of 5 cm water and peak inspiratory pressure of 9 cm of water). Inspiratory time of one second and respiratory rate of 30/min will always be maintained.
  * The infant will then receive a mean airway pressure of 5 cm water (positive end expiratory pressure of 4 cm water and peak inspiratory pressure of 6 cm of water).
  Interventions: Device: n-BiPAP
- NIPPV (Active Comparator): o The NIPPV group will receive at extubation a positive end expiratory pressure of 5 cm water, peak inspiratory pressure of 15cm of water, RRof35 and Ti of 0.32
  Interventions: Device: NIPPV

INTERVENTIONS:
Device: N-CPAP — The n-CPAP group will receive at extubation a single level continuous positive airway pressure of 7 cm water for at least 48 hours before weaning is commenced. If the infant is stable for the preceding 48 hours defined by having fewer than three minor apneas and no increase in oxygen requirement, weaning will be permitted.
  CPAP will be decreased from 6 cm water by 1 cm water every 24 hours if tolerated based on the above criteria. This will be done until a pressure of 4 cm water is reached.
  If a pressure of 4 cm water is successfully tolerated for 48 hours then time off n-CPAP will be allowed. Thereafter, no fixed weaning regime based on number of hours in a day the infant will be allowed to come off CPAP will be prescribed.
  Arms: n-CPAP
Device: n-BiPAP — The n-BiPAP group will receive at extubation a mean airway pressure of 7 cm water (positive end expiratory pressure of 5 cm water and peak inspiratory pressure of 9 cm of water). Inspiratory time of one second and respiratory rate of 30/min will always be maintained.
  The infant will then receive a mean airway pressure of 5 cm water (positive end expiratory pressure of 4 cm water and peak inspiratory pressure of 6 cm of water).
  Arms: n-BiPAP
Device: NIPPV — The NIPPV group will receive at extubation a positive end expiratory pressure of 5 cm water , a peak inspiratory pressure of 9 cm of water, RR of 35 and ti of 0.32
  Arms: NIPPV

SUMMARY:
non-invasive ventilation in preterms complaining from RDS a randomized, controlled trial to compare between capap, n-bipap and NIPPV

DETAILED DESCRIPTION:
The primary aim of this study is to compare the impact of early extubation to nasal continuous positive airway pressure (n-CPAP) versus nasal Bilevel positive airway pressure (n-BiPAP) and non invasive positive pressure ventilation(NIPPV) on the need for mechanical ventilation via endotracheal tube (MVET) to 7 days of age or less in preterm infants less than or equal to 34 weeks' gestation requiring intubation and surfactant if indicated for respiratory distress syndrome within 120 min of delivery . Second aim is to compare different outcomes of post-extubation n-CPAP , n-BiPAPand NIPPV.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants lessthan 34wk

Exclusion Criteria:

* preterms less than 1000 g birth weight
* infants with apgar 0at 1 min
* presenceofany other cause of respiratory distress as: congenital malformation affecting the cardiorespiratory system ,neuromuscular disease ,fetal hydrops , interventricular hemorrhage and chromosomal aberrations

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Failure of extubation during the first 48 hours post-extubation | during the first 48 hours post-extubation
  This will be defined as:
  1. Uncompensated respiratory acidosis defined as pH less than 7.2 and partial pressure of carbon dioxide of more than 60 mmHg (or)
  2. Major apnea requiring mask ventilation

SECONDARY OUTCOMES:
total days of non invasive ventilation | for 10 days from the hour of extubation
  anytime requiring respiratory support during a 24 hour clock counted as a day
length of hospital stay | 30 days postnatal age
  time of total admission
pneumothorax | 10 days post extubation
  air leak detected and was evident in chest x ray

CONTACTS AND LOCATIONS:
Overall Officials: Rania EL-Farrash, MD, Principal Investigator — Professor of paediatrics Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt